CLINICAL TRIAL: NCT05728970
Title: A Prospective Multicenter Study Conducted to Evaluate the Performance of the LumiraDX SARS-CoV-2 Ag Ultra and LumiraDX SARS-CoV-2 & Flu A/B Tests at Point of Care Sites
Brief Title: Performance Evaluation of the LumiraDX SARS-CoV-2 Ag Ultra and LumiraDX SARS-CoV-2 & Flu A/B Tests at Point of Care (POC) Sites
Acronym: PURSUE
Status: Completed | Type: Observational
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: S-CLIN-PROT-00056
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: SARS-CoV-2; Influenza A; Influenza B; COVID-19
Keywords: LumiraDx; Diagnostic tests; Multiplex; SARS-CoV-2; Influenza A; Influenza B; COVID-19; Infections; Coronavirus; Lung disease
MeSH Terms: conditions — COVID-19; Infections; Coronavirus Infections; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal and nasopharyngeal swab samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- symptomatic: Self-reported symptoms by the subject and/or preliminary assessment of the subject by the Investigator/designee should be suggestive of COVID-19 and/or Influenza at the time of the study visit. The subject must present as symptomatic, exhibiting one or more of the following signs and symptoms: fever, cough, shortness of breath, difficulty breathing, muscle pain, headache, sore throat, chills, repeated shaking with chills, new loss of taste or smell congestion or runny nose, diarrhea, nausea or vomiting. The onset of these symptoms will be recorded and will be within the last twelve (12) days
  Interventions: Diagnostic Test: LumiraDx SARS-CoV-2 Ag Ultra; Diagnostic Test: LumiraDx SARS-CoV-2 & Flu A/B

INTERVENTIONS:
Diagnostic Test: LumiraDx SARS-CoV-2 Ag Ultra — The LumiraDx SARS-CoV-2 Ag Ultra Test is an automated rapid microfluidic immunofluorescence assay for use with the LumiraDx Platform intended for the qualitative detection of the nucleocapsid protein antigen to SARS-CoV-2 directly from anterior nasal swab samples collected from symptomatic individuals within the first twelve days of symptom onset suspected of COVID-19 by their healthcare provider.
Diagnostic Test: LumiraDx SARS-CoV-2 & Flu A/B — The LumiraDx SARS-CoV-2 & Flu A/B test is an automated rapid microfluidic immunofluorescence assay for use with the LumiraDx Platform, for near-patient testing, intended for the qualitative detection and differentiation of SARS-CoV-2, Influenza A and/or Influenza B viral antigens from nasal swab samples.

SUMMARY:
This is a prospective multicenter study conducted to evaluate the performance of the LumiraDx SARS-CoV-2 Ag Ultra test in detecting severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and LumiraDx SARS-CoV-2 & Flu A/B test in differential detection of SARS-CoV-2, Influenza A (Flu A) and Influenza B (Flu B) at point of care sites. Subjects presenting with symptoms suggestive of coronavirus disease 2019 (COVID-19) and/or Influenza at the time of the study visit will be enrolled and asked to donate swab sample(s) for testing in the device(s) under evaluation.

DETAILED DESCRIPTION:
Approximately two thousand (2000) subjects will be enrolled in this study. Patients presenting to the study sites that meet the eligibility criteria will be considered for the study.

A subject's participation in this study will consist of a single on-site visit. Following completion of the informed consent process and a review of inclusion/exclusion criteria to determine eligibility, each subject will receive a unique study identification number.

Specimens will be obtained from each subject enrolled using standard collection methods.

The objectives of this study are to evaluate and validate the performance of:

* LumiraDx SARS-CoV-2 Ag Ultra test in detecting SARS-CoV-2 from symptomatic patients as compared with a Food and Drug Administration (FDA) cleared reverse transcription-polymerase chain reaction (RT-PCR) test.
* LumiraDx SARS-CoV-2 & Flu A/B tests in detecting SARS-CoV-2, Flu A, and/or Flu B from symptomatic patients as compared with an FDA cleared RT-PCR test for SARS-CoV-2 and an FDA cleared RT-PCR test for Flu A and Flu B.

ELIGIBILITY:
Inclusion Criteria:

1. Subject may be of any age or sex.
2. Self-reported symptoms by the subject and/or preliminary assessment of the subject by the Investigator/designee should be suggestive of COVID-19 and/or Influenza at the time of the study visit. The subject must present as symptomatic, exhibiting one or more of the following signs and symptoms: fever, cough, shortness of breath, difficulty breathing, muscle pain, headache, sore throat, chills, repeated shaking with chills, new loss of taste or smell congestion or runny nose, diarrhea, nausea or vomiting. The onset of these symptoms will be recorded and will be within the last twelve (12) days.
3. Participant (or parent/legal guardian) capable and willing to give informed consent/assent.

Exclusion Criteria:

1. The subject underwent a nasal wash/aspirate as part of standard of care testing during this study visit.
2. The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
3. Subjects undergoing treatment currently and/or within the past thirty (30) days of the study with medication to treat novel Coronavirus SARS-CoV-2 viral infections, which may include but is not limited to; COVID-19 antivirals (Lagevrio, PAXLOVID), Remdesivir (Veklury) or receiving convalescent plasma therapy for SARS-CoV-2.
4. Subjects undergoing treatment currently and/or within the past fourteen (14) days of the study visit with an inhaled influenza vaccine (FluMist®) or with anti-viral medication, which may include but is not limited to Amantadine (Symmetrel®), Rimantadine (Flumadine®), Zanamivir (Relenza®), Oseltamivir (Tamiflu®), Baloxavir Marboxil (Xofluza™), Palivizumab (Synagis®), or ribavirin.
5. The subject previously participated in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The entire population that met the inclusion criteria and none of the exclusion criteria. Symptomatic subjects will have symptoms suggestive of COVID-19 and/or Influenza.
Sampling Method: Non-Probability Sample
Enrollment: 716 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Performance evaluation of the LumiraDx SARS-CoV-2 Ag Ultra by health care professionals | 6 months
  Evaluate the performance of the LumiraDx SARS-CoV-2 Ag Ultra test in detecting SARS-CoV-2 in fresh nasal swab specimens from symptomatic patients. Performance will be evaluated by use of statistical analysis techniques to assess sensitivity (true positive rate), specificity (true negative rate), Negative and Positive Percent Agreement (NPA, PPA) of the LumiraDx test results versus an FDA-approved method where a result of 100% sensitivity, specificity, NPA or PPA would equate to complete agreement with the reference method and 0% would equate to no agreement.
Performance evaluation by health care professionals | 6 months
  Evaluate the performance of the LumiraDx SARS-CoV-2 & Flu A/B test in detecting and differentiating SARS-CoV-2, influenza A and influenza B in fresh nasal swab specimens from symptomatic patients. Performance will be evaluated by use of statistical analysis techniques to assess sensitivity (true positive rate), specificity (true negative rate), Negative and Positive Percent Agreement (NPA, PPA) of the LumiraDx test results versus an FDA-approved method where a result of 100% sensitivity, specificity, NPA or PPA would equate to complete agreement with the reference method and 0% would equate to no agreement.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Paragon Rx Clinical, Inc, Garden Grove, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Hillcrest Medical Research, LLC, DeLand, Florida
  - Hillcrest Medical Research, DeLand, Florida
  - Marisela Gonzalez MD PA, Miami, Florida
  - Barrett Clinic, La Vista, Nebraska
  - Meridian Clinical Research, Lincoln, Nebraska
  - Mercy Family Clinic, Dallas, Texas
  - Alliance for Multispecialty Research, LLC, Layton, Utah
  - Meridian Clinical Research, LLC. / Velocity Clinical Research, Hampton, Virginia